CLINICAL TRIAL: NCT02109822
Title: Pilot Observational Study to Determine Feasibility of a Standardized Treatment of Pulmonary Exacerbations in Patients With Cystic Fibrosis
Brief Title: Pilot Observational Study to Determine Feasibility of a Standardized Treatment of Pulmonary Exacerb. in Patients With CF
Acronym: STOP-OB-13
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Medical University of South Carolina (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Chris Goss, Professor of Medicine, University of Washington
Other Study IDs: 46256-EA
Record Dates: First submitted 2014-03-06; First posted 2014-04-10 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Cystic Fibrosis; Lung Infection; Cystic Fibrosis Pulmonary Exacerbation
Keywords: Cystic Fibrosis; Pulmonary Exacerbation; Lung Infection; Cystic Fibrosis Foundation; Cystic Fibrosis Foundation National Patient Registry
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CF patients with pulmonary exacerbations: Patients with CF who are hospitalized with a pulmonary exacerbation treated with intravenous antibiotics.

SUMMARY:
The goal of this research study is to better understand current treatment practices for pulmonary exacerbations (lung infections) and whether the Cystic Fibrosis National Patient Registry (CFFNPR)can be used for this type of study.

DETAILED DESCRIPTION:
Cystic fibrosis (CF), a life-shortening genetic disease, is marked by acute episodes during which symptoms of lung infection increase and lung function decreases. These pulmonary exacerbations (PEs) are treated with varying antibiotics for varying time periods based on needs determined by individual patients, their families, and the health care providers. Cystic fibrosis pulmonary guidelines for the treatment of PE published by the Cystic Fibrosis Foundation (CFF) in 2009 provided recommendations for treatment and also identified key questions for which additional studies were needed.

Standard treatment for PE involves many facets including selection of antibiotics, duration of use, and outcomes that define treatment success. Understanding current treatment practices and measures of treatment success are needed before a study can be designed to define optimal treatment strategies.

This is a multi-center, prospective, observational study designed to prospectively follow patients with CF that are initially admitted to the hospital for treatment of a pulmonary exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥12 years of age at Visit 1
* Enrolled in the CFFNPR (Patients may enroll in the Registry at Visit 1 if not previously enrolled.)
* Current hospitalization for treatment of a pulmonary exacerbation
* Planned hospital admission of at least 5 days with intravenous (IV) antibiotics at Visit 1
* Able to perform spirometry at admission and willing to perform spirometry on subsequent treatment and visit days
* Willing and able to complete symptom score daily
* Willing to return for a follow up visit at end of treatment (if necessary) and 28 days after start of IV antibiotic therapy
* Written informed consent (and assent when applicable) obtained from the participant or participant's legal representative

Exclusion Criteria:

* Previous enrollment in this study
* Treatment with IV antibiotics in the 6 weeks prior to Visit 1
* Admission to the intensive care unit for current pulmonary exacerbation
* Pneumothorax on admission
* Current hospitalization for scheduled pulmonary clean out
* Current hospitalization for sinusitis as the primary diagnosis
* Massive hemoptysis defined as > 250 cc in a 24 hour period, or 100 cc/day over 4 consecutive days occurring within one week of Visit 1
* Current pulmonary exacerbation thought to be due to allergic bronchopulmonary aspergillosis (ABPA)
* Ongoing treatment with prednisone equivalent >10 mg/day for greater than 2 weeks initiated prior to Visit 1
* History of solid organ transplantation Currently receiving antimicrobial therapy to treat non-tuberculous mycobacterium (e.g., M. abscessus, M. avium complex)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Cystic Fibrosis who are hospitalized with a pulmonary exacerbation treated with intravenous antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of using the CFF National Patient Registry | 28 days from time of start of IV antibiotic therapy.
  Assess feasibility using the CFF National Patient Registry as measured by the accuracy of data entry

SECONDARY OUTCOMES:
Physician and patient level clinical outcomes for their use in comparative studies of CF pulmonary exacerbations to determine the optimal treatment endpoints | During hospitalization and during a period following discharge of 28 days from time of start of IV antibiotic therapy.
  Evaluate physician assessment of treatment response as measured by the physician treatment assessment questionnaire. Evaluate change in lung function and patient reported respiratory symptoms and quality of life in response to treatment of an acute pulmonary exacerbation.

OTHER OUTCOMES:
Variability of practicing clinicians' treatment objectives, approaches, and assessment of outcomes related to CF pulmonary exacerbation | during hospitalization and during a period following discharge of 28 days from time of start of IV antibiotic therapy.
  Describe the variability of practicing clinicians' treatment objectives as measured by the physician assessment questionnaire, treatment approaches as measured by the choices of medications (specifically antibiotics), and assessment of patient level outcomes related to CF pulmonary exacerbation (change in lung function as measured by spirometry, respiratory symptoms as measure by the CFRSD-CRISS questionnaire) and health related quality of life (as measured by the EQ-5D questionnaire).
Inform the design of future pragmatic research of CF pulmonary exacerbation | During hospitalization and during a period following discharge of 28 days from time of start of IV antibiotic therapy.
  Identify the appropriate target patient population for future clinical trials by clarifying required stratification factors, and estimating target treatment effects and variability of treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H. Goss, MD MSc, Principal Investigator — University of Washington; Patrick Flume, MD, Principal Investigator — Medical University of South Carolina
Locations (12):
- United States (12):
  - CFF Adult Program University of Alabama, Birmingham, Alabama
  - CFF Care Center Arizona Health Science Center, Tucson, Arizona
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins, Baltimore, Maryland
  - CFF Care Center & Pediatric Program Rainbow Babies and Children's Hospita, Cleveland, Ohio
  - Rainbow Babies and Children's Hospital & University Hospitals Case Medical Center, Cleveland, Ohio
  - CFF Care Center & Pediatric Program Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CFF Care Center & Pediatric Program The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - CFF Care Center & Pediatric Program Seattle Children's Hospital, Seattle, Washington
  - University of Washington, Seattle, Washington
  - CFF Care Center & Pediatric Program University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data will be available once the primary manuscripts are published. Data without identifiers will be available through the Cystic Fibrosis Therapeutics Development Network Coordinating Center once an application to use the data is approved.

REFERENCES:
- [Derived] VanDevanter DR, Heltshe SL, Sanders DB, West NE, Skalland M, Flume PA, Goss CH; STOP-OB Study. Changes in symptom scores as a potential clinical endpoint for studies of cystic fibrosis pulmonary exacerbation treatment. J Cyst Fibros. 2021 Jan;20(1):36-38. doi: 10.1016/j.jcf.2020.08.006. Epub 2020 Aug 13. PMID 32800708
- [Derived] Stuart Elborn J, Geller DE, Conrad D, Aaron SD, Smyth AR, Fischer R, Kerem E, Bell SC, Loutit JS, Dudley MN, Morgan EE, VanDevanter DR, Flume PA. A phase 3, open-label, randomized trial to evaluate the safety and efficacy of levofloxacin inhalation solution (APT-1026) versus tobramycin inhalation solution in stable cystic fibrosis patients. J Cyst Fibros. 2015 Jul;14(4):507-14. doi: 10.1016/j.jcf.2014.12.013. Epub 2015 Jan 13. PMID 25592656